CLINICAL TRIAL: NCT05883449
Title: A Phase 2, Open-Label, Multi-Center Study of Innate Cell Engager AFM13 in Combination With Allogeneic Natural Killer Cells (AB-101) in Subjects With Recurrent or Refractory Hodgkin Lymphoma and CD-30 Positive Peripheral T-Cell Lymphoma
Brief Title: Phase 2 Study of AFM13 in Combination With AB-101 in Subjects With R/R HL and CD30+ PTCL
Acronym: LuminICE-203
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to sponsor decision
Sponsor: Affimed GmbH (Industry)
Collaborators: Artiva Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AFM13-203
Record Dates: First submitted 2023-05-19; First posted 2023-06-01 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Relapsed or Refractory Hodgkin Lymphoma; Peripheral T Cell Lymphoma
MeSH Terms: conditions — Recurrence; Hodgkin Disease; Lymphoma, T-Cell, Peripheral | interventions — AFM13; Cyclophosphamide; fludarabine; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Safety run-in in Hodgkin Lymphoma (Experimental): 4 safety run-in cohorts:
  * Cohort 1: 200 mg AFM13 + AB-101 (2 × 10e9 cells on Day 1, Day 8, Day 15)
  * Cohort 2: 300 mg AFM13 + AB-101 (2 × 10e9 cells on Day 1, Day 8, Day 15)
  * Cohort 3: 200 mg AFM13 + AB-101 (4 × 10e9 cells on Day 1; 2 × 10e9 cells on Day 8, Day 15)
  * Cohort 4: 300 mg AFM13 + AB-101 (4 × 10e9 cells on Day 1; 2 × 10e9 cells on Day 8, Day 15)
  Interventions: Drug: AFM13; Drug: AB-101; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Interleukin-2
- Dose Level A in Hodgkin Lymphoma (Experimental): Randomized Simon 2-stage design in Hodgkin Lymphoma Dose Level A (selected from cohort 1-4 of Safety run-in)
  Interventions: Drug: AFM13; Drug: AB-101; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Interleukin-2
- Dose Level B in Hodgkin Lymphoma (Experimental): Randomized Simon 2-stage design in Hodgkin Lymphoma Dose Level B (selected from cohort 1-4 of Safety run-in)
  Interventions: Drug: AFM13; Drug: AB-101; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Interleukin-2
- Exploratory: AFM13 + AB-101 on CD30-positive PTCL (Experimental): AFM13 + AB-101 on select CD30-positive PTCL subtypes (Dose Level A or B)
  Interventions: Drug: AFM13; Drug: AB-101; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Interleukin-2

INTERVENTIONS:
Drug: AFM13 — anti-human CD30 × anti-human CD16A recombinant antibody therapy, intravenous infusion
Drug: AB-101 — NK cell therapy, intravenous infusion
Drug: Cyclophosphamide — Lymphodepleting chemotherapy, intravenous infusion
Drug: Fludarabine — Lymphodepleting chemotherapy, intravenous infusion
Drug: Interleukin-2 — Immune cytokine, subcutaneously

SUMMARY:
AFM13-203 is a phase 2, open-label, multi-center, multi-cohort study with a safety run-in followed by expansion cohorts. The study is evaluating the safety and efficacy of AFM13 in combination with AB-101 in subjects with R/R classical HL and CD30-positive PTCL.

DETAILED DESCRIPTION:
The study will start with a safety run-in exploring AFM13/AB-101 combination treatment in subjects with classical HL. Two dose levels of AFM13 and AB-101, respectively, will be tested in 4 cohorts. Cohort 1 and 2 will enroll in parallel. Enrolment into Cohort 3 and 4 will start only if the combination treatment has been well tolerated.

Following the safety run-in observation period, a thorough risk-benefit analysis will be performed to determine 2 of the 4 cohorts/dose levels that will be further evaluated in the main part of the study which will also include subjects with classical HL and will follow a Simon two-stage design.

An additional exploratory cohort (Cohort 5) will enroll subjects with select CD30-positive PTCL subtypes after completion of the safety run-in.

All subjects will be treated with AFM13/AB-101 for a maximum of 3 cycles (cycle length is 48-days).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of FDG-avid relapsed or refractory classical HL OR select subtypes of FDG-avid CD30-positive relapsed or refractory PTCL
* For subjects with R/R PTCL a pre-enrollment tumor biopsy positive for CD30 locally assessed by Ber-H2 targeted immunohistochemistry at ≥1% is mandatory (PTCL subtypes: PTCL-NOS, Angioimmunoblastic T-cell lymphoma, ALCL, anaplastic lymphoma kinase (ALK)-positive, ALCL, ALK-negative)
* Subjects with R/R classical HL must have received at least two lines of therapy including one prior line of combination chemotherapy. Prior therapy must also have included brentuximab vedotin and a PD1 check point inhibitor.
* Subjects with R/R PTCL must have received at least one prior line of combination chemotherapy. Subjects with ALCL subtype of PTCL must have received or been intolerant to brentuximab vedotin.
* Subjects with R/R classical HL AND R/R PTCL: Prior ASCT is permitted if completed at least 3 months prior to the first dose of study treatment. Prior allogeneic stem cell transplantation will be permitted if completed at least 1 year from study enrollment and there are no signs or symptoms of GVHD. Prior CAR-T therapy is permitted if last CAR-T dose completed at least 6 months prior to the first dose of study treatment.
* Ability to understand and sign the ICF

Exclusion Criteria:

* Active central nervous system (CNS) involvement (untreated or uncontrolled parenchymal brain metastasis or positive cytology of cerebrospinal fluid)
* Previous treatment with AFM13 or CBNK cells
* History of a solid organ allograft, or an inflammatory or autoimmune disease likely to be exacerbated by IL-2 (including subjects requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease that may require systemic steroids or immunosuppressive agents
* Treatment with any therapeutic mAb or immunosuppressive medications
* Known active Hepatitis B or C defined per protocol
* Active HIV Infection
* History of any other systemic malignancy, unless previously treated with curative intent and the subject has been disease free for 2 years or longer
* Active acute or chronic graft vs. host disease (GVHD) or GVHD requiring immunosuppressive treatment, clinically significant central nervous system (CNS) dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2025-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wunderle Lydia, MD, Study Director — Affimed Inc.
Locations (15):
- United States (15):
  - O'Neal Comprehensive Cancer Center at UAB, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - UC Irvine Health, Orange, California
  - Sarah Cannon Research Institute, Denver, Colorado
  - Norton Cancer Institute, Louisville, Kentucky
  - Beth Israel Deaconess Medical, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UNC Immunotherapy Team, University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The three experimental Arms/Groups: 'Dose Level A in Hodgin Lymphoma', 'Dose Level B in Hodgin Lymphoma' and 'Exploratory: AFM13 + AB-101 on CD30-positive PTCL' were not enrolled due to the decision to terminate this study earlier, which was based solely on the financial situation of the company and was not related to the safety or efficacy.
Groups:
- Safety run-in Cohort 1: Cohort 1: 200 mg AFM13 + AB-101 (2 × 10e9 cells on Day 1, Day 8, Day 15)
  AFM13: anti-human CD30 × anti-human CD16A recombinant antibody therapy, intravenous infusion
  AB-101: NK cell therapy, intravenous infusion
  Cyclophosphamide: Lymphodepleting chemotherapy, intravenous infusion
  Fludarabine: Lymphodepleting chemotherapy, intravenous infusion
  Interleukin-2: Immune cytokine, subcutaneously
- Safety run-in Cohort 2: Cohort 2: 300 mg AFM13 + AB-101 (2 × 10e9 cells on Day 1, Day 8, Day 15)
  AFM13: anti-human CD30 × anti-human CD16A recombinant antibody therapy, intravenous infusion
  AB-101: NK cell therapy, intravenous infusion
  Cyclophosphamide: Lymphodepleting chemotherapy, intravenous infusion
  Fludarabine: Lymphodepleting chemotherapy, intravenous infusion
  Interleukin-2: Immune cytokine, subcutaneously
- Safety run-in Cohort 3: Cohort 3: 200 mg AFM13 + AB-101 (4 × 10e9 cells on Day 1; 2 × 10e9 cells on Day 8, Day 15)
  AFM13: anti-human CD30 × anti-human CD16A recombinant antibody therapy, intravenous infusion
  AB-101: NK cell therapy, intravenous infusion
  Cyclophosphamide: Lymphodepleting chemotherapy, intravenous infusion
  Fludarabine: Lymphodepleting chemotherapy, intravenous infusion
  Interleukin-2: Immune cytokine, subcutaneously
- Safety run-in Cohort 4: Cohort 4: 300 mg AFM13 + AB-101 (4 × 10e9 cells on Day 1; 2 × 10e9 cells on Day 8, Day 15)
  AFM13: anti-human CD30 × anti-human CD16A recombinant antibody therapy, intravenous infusion
  AB-101: NK cell therapy, intravenous infusion
  Cyclophosphamide: Lymphodepleting chemotherapy, intravenous infusion
  Fludarabine: Lymphodepleting chemotherapy, intravenous infusion
  Interleukin-2: Immune cytokine, subcutaneously
Period: Overall Study
Arm/Group | Safety run-in Cohort 1 | Safety run-in Cohort 2 | Safety run-in Cohort 3 | Safety run-in Cohort 4
Started | 6 | 7 | 6 | 6
Completed | 1 | 3 | 6 | 3
Not Completed | 5 | 4 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Safety run-in Cohort 1 | Safety run-in Cohort 2 | Safety run-in Cohort 3 | Safety run-in Cohort 4 | Total
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (20.68) | 43.6 (19.21) | 54.7 (14.61) | 46.0 (19.8) | 48.5 (18.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 4 | 4 | 17
  Male | 3 | 1 | 2 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 2
  White | 6 | 7 | 5 | 5 | 23
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 6 | 6 | 25

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) by Independent Radiology Committee
Description: Best ORR (complete response (CR) + partial response [PR]) by Independent Radiology Committee (IRC) based on positron emission tomography-computed tomography (PET-CT) as assessed by the Lugano classification. A participant will be assumed as a responder if he/she achieves complete or partial response at any postbaseline visit.
Time Frame: Disease assessments were conducted on Day 43 (+- 3 days) of each cycle. All subjects were treated for a maximum of 3 cycles.
Population: The Safety Run In Set (SRI) consists of all subjects of the 4 safety run-in cohorts who have received at least 66% of the combination dose during Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety run-in Cohort 1 | Safety run-in Cohort 2 | Safety run-in Cohort 3 | Safety run-in Cohort 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 5 | 5 | 6 | 5

2. Secondary Outcome: Duration of Response by Independent Radiology Committee
Description: Duration of response (DOR) defined as time from first assessment of PR or CR to the first assessment of progressive disease/death. Response based on positron emission tomography-computed tomography (PET-CT) as assessed by the Lugano classification assessed by Independent Radiology Committee.
Time Frame: Tumor assessment performed every 6 weeks for 3 cycles, if no disease progression on completion of treatment, then every 3 months for the first 12 months and then every 6 months (up to 20 months)
Population: All patients in the Safety Run In Set who had a response (CR or PR) assessed by the independent review committee.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Safety run-in Cohort 1 | Safety run-in Cohort 2 | Safety run-in Cohort 3 | Safety run-in Cohort 4
Number analyzed (Participants) | 5 | 5 | 6 | 5
months | 4.90 [2.20 to NA] — Not enough events to calculate the data | NA [NA to NA] — Not enough events to calculate the data | NA [NA to NA] — Not enough events to calculate the data | 6.97 [2.30 to NA] — Not enough events to calculate the data

3. Secondary Outcome: Complete Response Rate (CRR) by Independent Radiology Committee
Description: Complete Response Rate based on positron emission tomography-computed tomography (PET-CT) as assessed by the Lugano classification.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Safety run-in Cohort 1 | Safety run-in Cohort 2 | Safety run-in Cohort 3 | Safety run-in Cohort 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 4 | 3 | 4 | 3

4. Secondary Outcome: ORR by Investigator Based on PET-CT as Assessed by the Lugano Classification
Description: ORR (CR + PR) by Investigator based on positron emission tomography-computed tomography (PET-CT) as assessed by the Lugano classification
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Safety run-in Cohort 1 | Safety run-in Cohort 2 | Safety run-in Cohort 3 | Safety run-in Cohort 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 4 | 5 | 6 | 6

5. Secondary Outcome: Duration of Response by Investigator
Description: Duration of response (DOR) defined as time from first assessment of PR or CR to the first assessment of progressive disease/death. Response based on positron emission tomography-computed tomography (PET-CT) as assessed by the Lugano classification assessed locally by the Investigator.
Time Frame: as for outcome 2
Population: All patients in the Safety Run In Set who had a response (CR or PR) assessed by the investigator.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Safety run-in Cohort 1 | Safety run-in Cohort 2 | Safety run-in Cohort 3 | Safety run-in Cohort 4
Number analyzed (Participants) | 4 | 5 | 6 | 6
months | 3.86 [2.20 to NA] — Not enough events to calculate the data | 6.28 [2.10 to NA] — Not enough events to calculate the data | NA [NA to NA] — Not enough events to calculate the data | 4.65 [2.30 to NA] — Not enough events to calculate the data

6. Secondary Outcome: Incidence of Subjects Receiving Subsequent Transplant
Description: The number of subjects receiving subsequent transplant will be assessed and summarized by percentage rates
Time Frame: Throughout study completion (up to 20 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Safety run-in Cohort 1 | Safety run-in Cohort 2 | Safety run-in Cohort 3 | Safety run-in Cohort 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 1 | 2 | 0 | 1

7. Secondary Outcome: Frequency of Subjects With Study Drug Related TEAEs
Description: The number of subjects with study-drug related (AFM13 or AB-101) treatment-emergent adverse events (TEAEs)
Time Frame: From the time of first protocol-specific intervention until 30 days after the last administration (up to 20 months)
Population: The safety analysis set (SAS) will consist of all subjects who received any amount of any component of the regimen.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety run-in Cohort 1 | Safety run-in Cohort 2 | Safety run-in Cohort 3 | Safety run-in Cohort 4
Number analyzed (Participants) | 6 | 7 | 6 | 6
Participants | 5 | 4 | 5 | 5

8. Secondary Outcome: Frequency of Subjects With Serious Treatment Emergent Adverse Events
Description: The number of subjects who had serious treatment emergent adverse events.
Time Frame: From the time of first protocol-specific intervention until 30 days after the last administration (up to 20 months)
Population: The safety analysis set (SAS) will consist of all subjects who received any amount of any component of the regimen.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety run-in Cohort 1 | Safety run-in Cohort 2 | Safety run-in Cohort 3 | Safety run-in Cohort 4
Number analyzed (Participants) | 6 | 7 | 6 | 6
Participants | 2 | 5 | 4 | 5

9. Secondary Outcome: Frequency of Subjects Developing Anti-drug Antibodies (ADAs) Against AFM13
Description: The number of subjects developing anti-drug antibodies (ADAs) against AFM13
Time Frame: During treatment cycles (up to 6 months)
Population: The safety analysis set (SAS) will consist of all subjects who received any amount of any component of the regimen.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety run-in Cohort 1 | Safety run-in Cohort 2 | Safety run-in Cohort 3 | Safety run-in Cohort 4
Number analyzed (Participants) | 6 | 7 | 6 | 6
Participants | 2 | 1 | 2 | 1

10. Secondary Outcome: Progression-free Survival (PFS) by Independent Radiology Committee
Description: Progression-free survival (PFS) defined as time from first treatment (AFM13/AB-101) received until progressive disease (PD). Subjects who started a new anti-lymphoma therapy prior to a documented progressive disease were censored at the last disease assessment prior to initiation of new anti-lymphoma therapy. Subjects who discontinued the study before the first assessment of progressive disease or death were censored at their last disease assessment.
Time Frame: From the first treatment received until the first progression disease assessed by IRC or death.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Safety run-in Cohort 1 | Safety run-in Cohort 2 | Safety run-in Cohort 3 | Safety run-in Cohort 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
months | 4.17 [1.45 to NA] — Not enough events to calculate the data. | 7.66 [1.28 to NA] — Not enough events to calculate the data. | NA [NA to NA] — Not enough events to calculate the data. | 8.28 [1.35 to NA] — Not enough events to calculate the data.

11. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) was defined as (date of death - date of first dose)/30.4375. Patients alive at the end of study will be censored on the last date of observation.
Time Frame: From the first treatment received until the death.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Safety run-in Cohort 1 | Safety run-in Cohort 2 | Safety run-in Cohort 3 | Safety run-in Cohort 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
months | NA [NA to NA] — Not enough events to calculate the data. | 12.25 [3.48 to NA] — Not enough events to calculate the data. | 9.72 [NA to NA] — Not enough events to calculate the data. Due to high levels of participant censoring CI could not be calculated while median was able to be determined. | NA [NA to NA] — Not enough events to calculate the data.

ADVERSE EVENTS:
Time Frame: From the time of first protocol-specific intervention until 30 days after the last administration (up to 20 months)
Description: The safety analysis set (SAS) will consist of all subjects who received any amount of any component of the regimen.
Arm/Group | Safety run-in Cohort 1 | Safety run-in Cohort 2 | Safety run-in Cohort 3 | Safety run-in Cohort 4
All-Cause Mortality (participants affected / at risk) | 1/6 | 4/7 | 1/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6 | 5/7 | 4/6 | 5/6
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety run-in Cohort 1 (N=6) | Safety run-in Cohort 2 (N=7) | Safety run-in Cohort 3 (N=6) | Safety run-in Cohort 4 (N=6)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus Infection Reactivation (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus Oesophagitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus Viraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pseudomonas Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytokine Release Syndrome (Immune system disorders) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (3) | 0 (0) | 2 (5)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety run-in Cohort 1 (N=6) | Safety run-in Cohort 2 (N=7) | Safety run-in Cohort 3 (N=6) | Safety run-in Cohort 4 (N=6)
Nausea (Gastrointestinal disorders) | 5 (6) | 6 (14) | 4 (6) | 4 (6)
Constipation (Gastrointestinal disorders) | 4 (7) | 5 (8) | 3 (4) | 2 (3)
Vomiting (Gastrointestinal disorders) | 4 (10) | 5 (7) | 2 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 3 (3) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Oral Pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anal Fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal Incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oroantral Fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal Fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (5) | 5 (7) | 4 (5) | 1 (1) — General Disorders And Administration Site Conditions
Pyrexia (Gastrointestinal disorders) | 4 (6) | 5 (5) | 0 (0) | 2 (7) — General Disorders And Administration Site Conditions
Chills (General disorders) | 2 (6) | 4 (5) | 1 (2) | 2 (3) — General Disorders And Administration Site Conditions
Oedema Peripheral (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Injection Site Reaction (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Catheter Site Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza Like Illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection Site Induration (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (3) | 1 (1) | 3 (4) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 | 0 (0)
Rhinovirus Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cytomegalovirus Infection Reactivation (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis Infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterovirus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hcov-Oc43 Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral Herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parainfluenzae Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 2 (4) | 4 (22) | 4 (10) | 2 (4)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 3 (6) | 4 (7) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Brain Fog (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Extrapyramidal Disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle Spasticity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy Peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Restless Legs Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (12) | 2 (4) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (6) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure To Thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 3 (12) | 1 (4) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 1 (5) | 2 (7) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 2 (3) | 2 (4) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot Flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil Count Decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (5)
White Blood Cell Count Decreased (Investigations) | 0 (0) | 2 (4) | 0 (0) | 1 (2)
Platelet Count Decreased (Investigations) | 1 (1) | 0 (0) | 1 (5) | 0 (0)
Anti-Hla Antibody Test (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lipase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Protein Total Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Confusional State (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation Increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scleral Hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Strabismus (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytokine Release Syndrome (Immune system disorders) | 1 (2) | 0 (0) | 2 (4) | 0 (0)
Hypogammaglobulinaemia (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heavy Menstrual Bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The decision to terminate this study was based solely on the financial situation of the company and was not related to the safety or efficacy. Given this limitation, the results of the time to event endpoints are premature.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor has the right to review communications for 90 days prior to public release (whereby the sponsor may ask to consider modifications to ensure necessary protection of sponsor's IP). Any publication shall be not made before the first multi-centre publication if the study is a part of a multi-centred clinical trial. Also, if a publication concerns the analyses of data from a multi-centred clinical trial, the communication shall make reference to the relevant multi-centre publication

DOCUMENTS (2):
  • Study Protocol (2024-07-03): https://cdn.clinicaltrials.gov/large-docs/49/NCT05883449/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-23): https://cdn.clinicaltrials.gov/large-docs/49/NCT05883449/SAP_001.pdf